CLINICAL TRIAL: NCT07180602
Title: Healing Minds II: Biofeedback, Breathing Practices, Nutrition and Exercise Counseling in Children and Adolescents With ADHD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor cancelled the study before patients were enrolled.
Sponsor: Hoskinson Health and Wellness Clinic (Industry)
Responsible Party: Principal Investigator, Inara McMaster, Director of Pediatrics, Hoskinson Health and Wellness Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRANY IRB File #25-10-430-1498
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: Biofeedback; Nutrition Counseling; Exercise Counseling
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): One group, no-placebo comparer
  Interventions: Behavioral: Heart Math Biofeedback Breathing Practices; Behavioral: Nutrition Counseling combined with Exercise Counseling

INTERVENTIONS:
Behavioral: Heart Math Biofeedback Breathing Practices — Phase I and II (0-6 months): Biofeedback will be implemented based on the Heart Math Protocol. Breathing practices will include a variety of yoga and qi gong techniques.
Behavioral: Nutrition Counseling combined with Exercise Counseling — Phase II (3-6 months): Dietary education and an age-and gender-specific diet prescription based on the Mediterranean Diet. Nutrition counseling includes nutrition supplementation to correct deficiencies. Study participants will have a blood test to examine vitamins and minerals and identify deficiencies. Exercise counseling includes developmentally appropriate guidelines for cardiopulmonary, strength and flexibility activities based on guidelines from the ACSM and the AAP. Study participants and parents will be provided with a handout with exercise recommendations to follow at home and links to a website for additional suggestions for developmentally-appropriate physical activities and a tracking tool to assist parents with determining if their child is following the guidelines.

SUMMARY:
The Pediatric Healing Minds II intervention includes a biofeedback component, breathing practices nutrition and exercise counseling. Biofeedback is a type of mind-body technique used to control body functions such as heart, lung and muscle responses. Biofeedback uses therapeutic techniques that aim to help study participants gain more awareness and control over certain physiological functions in their bodies. It involves the use of electronic monitoring equipment to provide real-time information about physiological processes such as heart rate, HRV, coherence and muscle tension. This information is then provided back to the study participant, allowing them to learn how to consciously regulate these processes. During the sessions parents are expected to attend and participate. Study participants and parents will have access to a video that provides instructions for placement of the Heart Math single small ear lobe or finger sensor. Breathing Practices include alternate nostril, qi gong and other breathing practices. Nutrition counseling includes nutrition supplementation to correct deficiencies, dietary education and an age-and gender-specific diet prescription based on the Mediterranean Diet. Exercise counseling includes developmentally appropriate guidelines for cardiopulmonary, strength and flexibility activities based on guidelines from the American College of Sports Medicine (ACSM) and the American Academy of Pediatrics (AAP).

The objective of this research proposal is to examine the combined effects of an integrative approach including biofeedback, breathing practices, nutrition and exercise counseling intervention (Healing Minds II), on symptoms and severity of ADHD, impulsivity and attention (e.g., QB continuous performance test) in youth 7-18 years of age. The investigators hypothesize that ADHD symptoms and severity, impulsivity and attention will be significantly improved and coherence increased after participation in the 6-month intervention. The investigators also propose that ADHD severity in those patients with prescribed medication but poorly-controlled ADHD will demonstrate the greatest improvement compared to those not prescribed medication and those who have well-controlled ADHD.

DETAILED DESCRIPTION:
Attention-Deficit Hyperactivity Disorder (ADHD) affects 2.8% of adults and 5.9% of youth worldwide, and is more prevalent in males compared to females. There are both genetic and environmental risks for developing ADHD. As such, the condition is an epigenetic disorder with a complex pathophysiology that includes numerous biological pathways. Numerous co-morbidities are associated with ADHD including obesity, asthma, diabetes mellitus, and somatic disorders. Individuals diagnosed with ADHD are more likely to attempt and complete a suicide attempt. Chronic illnesses associated with ADHD are shown to develop early in life and track into adulthood. Thus, ADHD is a significant public health issue.

The diagnosis of ADHD is based on a standard criterion for validity of a mental disorder. A licensed clinician interviews the parent or guardian and/or patient and documents the established criteria for the disorder. There is a growing body of literature linking ADHD with other mental health disorders. Numerous studies report strong correlations between ADHD and trauma-related disorders such as post-traumatic stress disorder (PTSD), a serious psychological and physical illness with chronic health consequences including the development of additional mental disorders. Individuals diagnosed with PTSD experience traumatic life events that lead to a biological stress reaction, which negatively affect their overall emotional and mental health. Symptoms of PTSD include intrusions (involuntary and stressful memories of the trauma), avoidance of the trauma associated stimuli, and persistent physiological hyperarousal. These symptoms parallel those of ADHD, especially hyper arousal. Thus, interventions targeting multiple psychobiological pathways may improve the severity of ADHD.

Medications are often prescribed for the treatment of ADHD in youth; although, side effects limit their utility. Other treatment options for ADHD and related conditions in children and adolescents include cognitive-behavioral trauma-focused therapies and complementary, pharmacological therapy and alternative and integrative interventions.The latter of these is emerging as not only an enhancement to more traditional therapies, but as a viable replacement with promising treatment results. One such therapy, Biofeedback promotes the acquisition of psychophysiological self-regulation skills through the use of an operant conditioning procedure. Visual, auditory and tactile feedback is provided in real time to the participant in an effort to promote voluntary control over involuntary physiological processes, such as HRV and coherence. Increases in HRV and coherence are shown to positively impact anxiety, PTSD, and other measures of psychosocial well-being. However, there is limited evidence that biofeedback reduces ADHD symptomology in children and adolescents. Notably, the implementation of breathing practices in complementary and alternative interventions in children with ADHD is becoming increasingly popular among parents. This may be due to emerging research indicating that breathing practices may reduce stress and anxiety in adults and children. The Mediterranean Diet is shown to be associated with a lower risk of ADHD and other mental health disorders in children and adolescents. Recent research also demonstrates that the Mediterranean diet improves ADHD symptoms in youth. Participation in exercise including aerobic activities is also shown to improve ADHD symptoms in children and adolescents. However, the effect of breathing practices in combination with biofeedback, nutrition and exercise on ADHD symptoms and severity, impulsivity and attention in youth with ADHD is unknown.

Intervention Methods: The study participant will attend sessions weekly during Phase I and monthly during Phase II of the intervention at the Hoskinson Health and Wellness Clinic. The parent(s) or guardian will accompany the study participant and follow along with the cues during the weekly session. Prior research indicates that parenting behaviors are important determinants in modifying symptoms in youth with ADHD. Each session will be approximately 60 minutes. The principal investigator/pediatrician or trained and certified health care or research staff member will deliver the intervention. Biofeedback will be implemented based on the Heart Math Protocol. Breathing practices will include a variety of yoga and qi gong techniques. Nutrition counseling includes nutrition supplementation to correct deficiencies, dietary education and an age-and gender-specific diet prescription based on the Mediterranean Diet. Exercise counseling includes developmentally appropriate guidelines for cardiopulmonary, strength and flexibility activities based on guidelines from ACSM and AAP.

The Pediatric Healing Minds II intervention includes a biofeedback component and breathing practices. Biofeedback is a type of mind-body technique used to control body functions such as heart, lung and muscle responses. Biofeedback uses therapeutic techniques that aim to help study participants gain more awareness and control over certain physiological functions in their bodies. It involves the use of electronic monitoring equipment to provide real-time information about physiological processes such as heart rate, heart rate variability, coherence and muscle tension. This information is then provided back to the study participant, allowing them to learn how to consciously regulate these processes. During the sessions parents are expected to attend and participate. Study participants and parents will have access to a video that provides instructions for placement of the Heart Math single small ear lobe or finger sensor. Breathing Practices include qi gong and other breathing practices.

Our specific aims are as follows:

AIM I. Conduct a one group, no-placebo comparer, pre-post observational clinical trial in children and adolescents 7-18 years of age diagnosed with ADHD (N=16) to examine the additive effects of:

* 20-weeks of an integrative intervention (Healing Minds II) that includes Heart Math Biofeedback Breathing Practices (Phase I and II; 0-6 months),
* 10 weeks of Nutrition Counseling combined with Exercise Counseling (Phase II; 3-6 months)

AIM Ia. Observe the effects of the Healing Minds II intervention in the following sub-groups of youth:

* ADHD without medication (well versus poorly controlled)
* ADHD with medication (well versus poorly controlled)

Assessment of Efficacy: Specifications of the efficacy parameters, which will be obtained during Day 1 of baseline and follow-up are below. Participants will receive coherence by ECG weekly during the Phase I and monthly during Phase II of intervention:

* Diagnosis of ADHD will be determined by the DSM-5-TR method using the Vanderbilts-PT
* Impulsivity and attention by QBTest
* Coherence by ECG according to the Heart Math protocol

All study measures will be obtained during the baseline visit, 1-4 weeks prior to the intervention, and the follow-up visits, 1-4 weeks post the Phase I intervention and 1-4 weeks post the Phase II intervention. The coherence by ECG assessment will be conducted weekly during Phase I and monthly during Phase II of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 7-18 years
* Male and female children and adolescents
* Confirmed diagnosis of ADHD using the DSM-5-TR criteria

Exclusion Criteria:

* Severe, uncontrolled mental illness including depression, panic disorders
* Suicidal ideology
* Psychosis
* Severe, uncontrolled, autonomic nervous system or metabolic disorders including hypertension, diabetes, hypotension, autoimmune disease, or any condition that would limit their participation in the intervention
* Disorders involving severe impairments of memory or neurological conditions such as seizures
* Pregnant or nursing females may not participate because of some of the tests that are required for the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ADHD Severity measured by DSM-5 method using the Vanderbilts-PT | Obtained during the baseline visit, and again at 3 and 6 months following the initiation of the intervention.
  Diagnosis of ADHD will be provided by the referring physician or performed by the study pediatrician based on the DSM-5-TR criteria using the - Vanderbilts-PT parent scales as per established clinical guidelines and procedures. Eighteen symptoms are rated on a scale of 0 to 3. The number of responses rated 2 (often) or 3 (very often) are totaled for inattentive symptoms (questions 1-9) and hyperactive symptoms (questions 10-18). Eight performance measures (questions 48-55) are rated on a scale of 1 to 5. The number of performance responses rated 4 (somewhat of a problem) or 5 (problematic) are totaled and an average performance score is calculated. A score of 6 out of 9 symptoms on questions 1-9 or from questions 10-18 PLUS a score of 4 or 5 on any of the performance questions indicate ADHD.
ADHD Severity measured by Impulsivity and Attention by QBTest | Obtained during the baseline visit, and again at 3 and 6 months following the initiation of the intervention.
  Impulsivity and attention will be determined by the QB continuous performance test (QB Test) using standard clinical procedures. QBTest is an objective ADHD test for children and adolescents 7-18 years. The test assesses impulsivity and attention using motion tracking using a computer-based system. Study participants will be presented with a series of target and non-target stimuli on a computer screen. The study physician, nurse or research staff member will instruct the study participant to select the target stimuli by pressing a button. They will be instructed to not press the button when a non-target stimulus is presented. The assessment will take approximately 15-20 minutes to complete. Data retrieved from the QBTest is analyzed using a comparative normative control group without ADHD. Each activity measure and impulse and control measure are given a Q-score and a percentile score as compared to the normative control group. Higher scores indicated ADHD.

SECONDARY OUTCOMES:
Coherence by ECG according to the Heart Math protocol | The coherence by ECG assessment will be conducted weekly during Phase I (0-3 months) and monthly during Phase II (3-6 months) of the intervention.
  Coherence by ECG will be assessed by the pediatrician or trained and certified health care or research staff member during weekly and monthly sessions using the Heart Math system according to established guidelines and procedures. An ear lobe and finger sensor will be provided for the (Heart Math) Biofeedback procedure and assessment. Fluctuations in the time interval between consecutive beats will be determined during the measurement of ECG as part of the Heart Math biofeedback standard protocol. The variation in the time interval between consecutive heartbeats, for each inter beat interval will be continuously recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Inara McMaster, MD, Principal Investigator — Hoskinson Health and Wellness Clinic
Locations (1):
- Hoskinson Health and Wellness Clinic, Gillette, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No